CLINICAL TRIAL: NCT03932344
Title: A Non-interventional, Post-authorization Safety Study (PASS) to Evaluate Long-term Safety of Anakinra (Kineret®) in Patients With Systemic Juvenile Idiopathic Arthritis
Brief Title: Long-term Safety Study of Kineret® in Patients With Systemic Juvenile Idiopathic Arthritis (SJIA)
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Anakin-302; ENCEPP/SDPP/28378 (Other: EU PAS register number)
Record Dates: First submitted 2019-04-16; First posted 2019-04-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Still Disease, Juvenile Onset
Keywords: SJIA; Kineret; Anakinra; Long term safety
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SJIA patients on Kineret treatment: SJIA patients on Kineret treatment enrolled in the Pharmachild JIA registry
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra according to prescription
  Other Names: Kineret

SUMMARY:
The purpose of the study is to evaluate and characterize long-term safety of Kineret when used in standard clinical practice to treat patients with systemic juvenile idiopathic arthritis (SJIA). The study will be based on already available data from the Pharmachild juvenile idiopathic arthritis (JIA) registry which holds the European Network of Centers for Pharmacoepidemiology and Pharmacovigilance (ENCePP) study seal.

DETAILED DESCRIPTION:
This is an international, non-interventional, single-armed, pharmacovigilance registry study on long-term safety of Kineret utilizing already available data from the ENCePP certified Pharmachild JIA registry.

The Paediatric Rheumatology International Trials Organisation (PRINTO) is a non-profit, non-governmental, international research network with the goal to foster, facilitate and co-ordinate the development, conduct, analysis, and reporting of multi-centers, international clinical trials and/or outcome standardization studies in children with paediatric rheumatic diseases.

The Pharmachild JIA registry, maintained by PRINTO, is a registry collecting data from patients with JIA including patients with SJIA. In the Pharmachild JIA registry 40 countries are participating of which 15 countries have collected data on Kineret treatment.

This study includes secondary use of data already available in the Pharmachild JIA registry.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a diagnosis of SJIA as per the International League of Associations for Rheumatology (ILAR) classification criteria
* Included in the Pharmachild registry
* Ever treated with Kineret subsequently to SJIA diagnosis

Exclusion Criteria:

No specific exclusion criteria will be applied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be extracted and analyzed for all male and female patients with a diagnosis of SJIA as per the ILAR classification criteria included in the Pharmachild registry and who were ever treated with Kineret subsequently to SJIA diagnosis. That is, all eligible patients participating in the Pharmachild JIA registry study are included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The occurrence of non-serious adverse events (AEs) of at least moderate severity and serious AEs (SAEs), including macrophage activation syndrome (MAS) as an event of special interest (ESI). | The Pharmachild registry was set up in December 2011. The first Kineret treatment, retrospectively collected in the registry, occurred in 2004. Data collected in the registry up until September 30, 2018 will be used (secondary use) in this study.
  The occurrence of non-serious AEs of at least moderate severity and serious AEs (SAEs), including MAS as an ESI. AEs (SAEs), including MAS as an ESI.
The duration of Kineret treatment in a real-world setting. | The Pharmachild registry was set up in December 2011. The first Kineret treatment, retrospectively collected in the registry, occurred in 2004. Data collected in the registry up until September 30, 2018 will be used (secondary use) in this study.
  The duration of Kineret treatment in a real-world setting.
The reasons for Kineret treatment discontinuation. | The Pharmachild registry was set up in December 2011. The first Kineret treatment, retrospectively collected in the registry, occurred in 2004. Data collected in the registry up until September 30, 2018 will be used (secondary use) in this study.
  The reasons for Kineret treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Swedish Orphan Biovitrum
Locations (1):
- IRCCS Istituto G. Gaslini, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Giancane G, Papa R, Vastert S, Bagnasco F, Swart JF, Quartier P, Anton J, Kamphuis S, Sanner H, Glerup M, De Benedetti F, Tsitsami E, Remesal A, Moreno E, De Inocencio J, Myrup C, Pallotti C, Kone-Paut I, Franck-Larsson K, Malmstrom H, Cederholm S, Pistorio A, Wulffraat N, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). Anakinra in Patients With Systemic Juvenile Idiopathic Arthritis: Long-term Safety From the Pharmachild Registry. J Rheumatol. 2022 Apr;49(4):398-407. doi: 10.3899/jrheum.210563. Epub 2022 Feb 1. PMID 35105709